CLINICAL TRIAL: NCT04670536
Title: The Degen Study: Post-market Clinical Follow-up on the PASS LP, PASS Degen and PASS Tulip Systems.
Brief Title: The Degen Study: Post-market Clinical Follow-up on the PASS LP, PASS Degen and PASS Tulip Systems (PASS DEGEN)
Acronym: PASS DEGEN
Status: Completed | Type: Observational
Sponsor: Medicrea International (Industry)
Responsible Party: Sponsor
Other Study IDs: 0313
Record Dates: First submitted 2020-12-03; First posted 2020-12-17 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Thoracolumbar Disc Degeneration; Thoracolumbar Spondylolisthesis; Spinal Deformity; Spinal Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- PASS LP implants: Patient suffering from a spinal degenerative disease and who is operated with PASS LP
  Interventions: Device: PASS LP implants
- PASS Degen implants: Patient suffering from a spinal degenerative disease and who is operated with PASS DEGEN
  Interventions: Device: PASS DEGEN
- PASS Tulip PRIME implants: Patient suffering from a spinal degenerative disease and who is operated with PASS TULIP PRIME
  Interventions: Device: PASS TULIP PRIME

INTERVENTIONS:
Device: PASS LP implants — Thoraco lumbar arthrodesis
  Groups: PASS LP implants
Device: PASS DEGEN — Thoraco lumbar arthrodesis
  Groups: PASS Degen implants
Device: PASS TULIP PRIME — Thoraco lumbar arthrodesis
  Groups: PASS Tulip PRIME implants

SUMMARY:
The purpose of this post-market clinical study is to evaluate the long-term safety and efficacy of the MEDICREA's systems PASS LP, PASS DEGEN, and PASS Tulip PRIME to treat degenerative diseases. This study is supporting the clinical evaluation report. From the standard-of-care perspective, the results of The Degen study are expected to contribute to a better understanding of expected safety and clinical outcomes from a short (intra- and peri-operative) to a medium-term follow-up (post-operatively).

ELIGIBILITY:
Inclusion Criteria:

* Patients of at least 18 years old
* Patient suffering from a spinal degenerative disease.
* Patient requiring spinal surgery for less than 4 levels for a spinal degenerative disease
* Patient implanted with MEDICREA's products, or patients who are candidate to receive including at least the PASS LP and/or PASS DEGEN and/or PASS TULIP Prime implants
* Patient affiliated to a national insurance system

Exclusion Criteria:

* Patient unable or unwilling to sign and understand an information note with proof of patient consent
* Patient unable to complete a self-administered questionnaire
* Patient presenting contra-indications to a Xray follow-up
* Patient of more than 18 years old under a protection procedure
* Patient judged as non-compliant by the investigator or not able to come back for follow-up visits up to 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Fusion | At 24months
  The primary endpoint is the fusion status of each patient at the 24-month visit postoperative. This fusion assessment will be done through the analysis of the standard of care imaging (CT-scan, X-rays, and/or MRI) by the investigator and through the clinical examination of the patient by the investigator.

SECONDARY OUTCOMES:
Evolution of the pain (VAS) | Preoperative, and 1-6, 12 and 24 months postoperative
  Change of leg and back pain score from the preoperative visit to all available postoperative timepoints: from 0 (better) to 10 (worst)
Quality of life with ODI | Preoperative, and 1-6, 12 and 24 months postoperative
  Change of non-validated ODI score from the preoperative visit to all available postoperative timepoints: from 0 (better) to 5 (worst)
Quality of life with SF-12 | Preoperative, and 1-6, 12 and 24 months postoperative
  Change of non-validated SF-12 score from the preoperative visit to all available postoperative timepoints: from to 0 (better) to 3 or 5 depending the question (worst)
Device or procedure-related adverse events and all SAEs up to 24 months | Preoperative, and 1-6, 12 and 24 months postoperative
  During the follow-up period, the occurrence of device and procedure related AEs and all serious adverse events will be monitored, registered, and analyzed. To safeguard the safety of the clinical study subjects, all SAEs will be collected even those that may not be directly related to the surgery.
Surgeons'satisfaction with these implants and instruments | During the surgery and until the 24months postoperative visit
  Surgeons will be requested to complete questions about device/surgery satisfaction.
Fusion status at the 1/6 month and 12-month visit | At the 1-6, and 12 months postoperative
  The primary objective is defined as the ability of the implant to promote the stabilization
Patient satisfaction at all available postoperative timepoints | At 1-6, 12 and 24 months postoperative
  Patient satisfaction is used to evaluate patient satisfaction after surgery and during the follow-up period.
  Satisfaction is measured at four different levels: 1 (better) to 4 (worst)

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique du Dos Bordeaux - Terrefort, Bruges
  - Clinique des Cèdres, Cornebarrieu
  - CHRU Tours, Hôpital de Bretonneau, Tours
  - Hôpital Pitié-Salpêtrière AP-HP, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Copay AG, Glassman SD, Subach BR, Berven S, Schuler TC, Carreon LY. Minimum clinically important difference in lumbar spine surgery patients: a choice of methods using the Oswestry Disability Index, Medical Outcomes Study questionnaire Short Form 36, and pain scales. Spine J. 2008 Nov-Dec;8(6):968-74. doi: 10.1016/j.spinee.2007.11.006. Epub 2008 Jan 16. PMID 18201937
- [Background] Hagg O, Fritzell P, Nordwall A; Swedish Lumbar Spine Study Group. The clinical importance of changes in outcome scores after treatment for chronic low back pain. Eur Spine J. 2003 Feb;12(1):12-20. doi: 10.1007/s00586-002-0464-0. Epub 2002 Oct 24. PMID 12592542
- [Background] Glassman SD, Carreon LY, Djurasovic M, Dimar JR, Johnson JR, Puno RM, Campbell MJ. Lumbar fusion outcomes stratified by specific diagnostic indication. Spine J. 2009 Jan-Feb;9(1):13-21. doi: 10.1016/j.spinee.2008.08.011. Epub 2008 Sep 19. PMID 18805059
- [Background] Fairbank JC. Why are there different versions of the Oswestry Disability Index? J Neurosurg Spine. 2014 Jan;20(1):83-6. doi: 10.3171/2013.9.SPINE13344. Epub 2013 Nov 8. PMID 24206036
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Johnsen LG, Hellum C, Nygaard OP, Storheim K, Brox JI, Rossvoll I, Leivseth G, Grotle M. Comparison of the SF6D, the EQ5D, and the oswestry disability index in patients with chronic low back pain and degenerative disc disease. BMC Musculoskelet Disord. 2013 Apr 26;14:148. doi: 10.1186/1471-2474-14-148. PMID 23622053
- [Background] Gum JL, Carreon LY, Stimac JD, Glassman SD. Predictors of Oswestry Disability Index worsening after lumbar fusion. Orthopedics. 2013 Apr;36(4):e478-83. doi: 10.3928/01477447-20130327-26. PMID 23590789
- [Background] Ghogawala Z, Whitmore RG, Watters WC 3rd, Sharan A, Mummaneni PV, Dailey AT, Choudhri TF, Eck JC, Groff MW, Wang JC, Resnick DK, Dhall SS, Kaiser MG. Guideline update for the performance of fusion procedures for degenerative disease of the lumbar spine. Part 3: assessment of economic outcome. J Neurosurg Spine. 2014 Jul;21(1):14-22. doi: 10.3171/2014.4.SPINE14259. PMID 24980580
- [Background] Gandek B, Ware JE, Aaronson NK, Apolone G, Bjorner JB, Brazier JE, Bullinger M, Kaasa S, Leplege A, Prieto L, Sullivan M. Cross-validation of item selection and scoring for the SF-12 Health Survey in nine countries: results from the IQOLA Project. International Quality of Life Assessment. J Clin Epidemiol. 1998 Nov;51(11):1171-8. doi: 10.1016/s0895-4356(98)00109-7. PMID 9817135